CLINICAL TRIAL: NCT01128868
Title: Treatment of Reverse Oblique Intertrochanteric or Subtrochanteric Fractures With a Proximal Femur Locking Compression Plate (PF-LCP, PF-LCP Hook Plate, PeriLoc) or Trochanteric Nails. A Multicenter Cohort Study
Brief Title: Proximal Femur Locking Compression Plates Versus Trochanteric Nails
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PF LCPs vs Trochanteric Nail
Record Dates: First submitted 2010-05-20; First posted 2010-05-24 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Reverse Oblique Intertrochanteric Fractures; Reverse Oblique Subtrochanteric Fractures
Keywords: Reverse oblique intertrochanteric fractures; Reverse oblique subtrochanteric fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Proximal femur locking plate (Active Comparator): Treatment of reverse oblique intertrochanteric or subtrochanteric fractures with a Proximal Femur Locking Compression Plate (PF-LCP, PF-LCP Hook Plate, PeriLoc)
  Interventions: Device: Proximal femur locking plate
- Trochanteric nail (Other): Treatment of reverse oblique intertrochanteric or subtrochanteric fractures with Trochanteric Nails (PFNA, TFN, GN)
  Interventions: Device: Intertrochanteric nail

INTERVENTIONS:
Device: Proximal femur locking plate — Proximal femur locking plate (PF-LCP, PF-LCP Hook Plate, Periloc)
  Other Names: LCP Proximal Femur Plate (Synthes); LCP Proximal Femur Hook Plate (Synthes); PeriLoc Periarticular Locked Plating System (Smith & Nephew)
  Arms: Proximal femur locking plate
Device: Intertrochanteric nail — Intertrochanteric nail (PFNA, TFN, GN)
  Other Names: Proximal Femoral Nail Antirotation (Synthes); Titanium Trochanteric Fixation Nail (Synthes); Gamma Trochanteric Nail (Stryker)
  Arms: Trochanteric nail

SUMMARY:
The purpose of this study is to compare the abductor muscle strength measured with a dynamometer in patients with reverse oblique inter- or subtrochanteric fractures treated either with a proximal femur locking plate or a trochanteric nail.

"Proximal femur locking plates" stands for both the PF-LCP (Synthes) and the PeriLoc (Smith & Nephew). Trochanteric nails allowed in this study are the Proximal Femoral Nail Antirotation (PFNA), the Titanium Trochanteric Fixation Nail (TFN) and the Gamma Nail (GN).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with closed or type 1 open reverse oblique intertrochanteric fractures (AO 31 - A3) or subtrochanteric fractures (transverse fracture line, main fracture line maximum 5 cm distal from the lesser trochanter; proximal extension of fracture allowed)
* Definitive fracture fixation with either a proximal femur locking plate or an intertrochanteric nail within 4 days after accident
* Signed written informed consent (by the subject or legal guardian) and agreement to attend the planned FUs
* Able to understand and read country national language at an elementary level

Exclusion Criteria:

* Pathologic fracture
* Polytrauma
* Any displacement of a femoral neck fracture
* Additional fracture of one of the lower extremities that significantly affects the functional outcome
* Additional injury of the lower limb that significantly affects the functional outcome
* Fractures of the upper extremity if it affects the mobility of the patient
* Type 2 or 3 open fracture
* Drug or alcohol abuse
* Active malignancy
* ASA class V and VI
* Inability to walk independently prior to injury
* Neurological and psychiatric disorders that would preclude reliable assessment
* Patient is not able to come to the regular FUs
* Patients who have participated in any other device or drug related clinical trial within the previous month
* Pregnancy (tested with a urine pregnancy test) or women planning to conceive within the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-05; Primary Completion 2013-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Compare the functional outcome and abductor muscle strength measured with Lafayette Manual Muscle Tester in patients with reverse oblique inter- or subtrochanteric fractures treated either with a proximal femur locking plate or a trochanteric nail. | one year
  As hip abductors are the most important muscles around the hip joint, the primary outcome parameter will involve objectively measuring hip abductor strength. Muscle strength will be assessed with a portable handheld dynamometer (Model 01163, Lafayette Instrument Company, Lafayette, IN, USA).

SECONDARY OUTCOMES:
Patient outcome | one year
  Patient outcome will be measured using the following outcome measurements:
  Mobility measured with the "timed up & go"-test (TUG), Lower Extremity Measure (LEM) for functional outcome, Length of hospital stay, Walking ability (Parker Mobility Score), Capacity to return to pre-residential status, Quality of life (Short Form-36 [SF-36]), Mortality.
Pain scores on the Visual Analog Scale | one year
  Pain will be measured with the Visual Analogue Scale (VAS) (additionally assessed in a subgroup with the Brief Pain Inventory [BPI]).
Patient satisfaction with the Visual Analogue Scale | one year
  Satisfaction measured with the VAS
Abductor muscle function with the Trendelenburg sign analysis | one year
  Abductor muscle function test
Surgical details | Initial hospitalization
  Skin-to-skin time, Fluoroscopy time, Blood loss, Blood transfusions, Surgeons experience.
Local complications | one year
  Local complication will be recorded and categorized:
  Implant / surgery complications, Bone / fracture complications, Soft tissue / wound complications.
Revision rate | one year
  Surgical revision includes all secondary surgical interventions that are related to the injury itself or the primary intervention. It is distinguished from planned revisions due to the injury (eg, planned soft tissue procedure) and revisions due to a complication. Revisions due to a complication are undertaken to resolve the problem and will therefore be documented in the complication form.
Systemic or general complications | one year
  All complications affecting other regions of the body will be documented and evaluated as general/systemic complications, eg, thromboembolic complications, sepsis and others.
Exploration of prognostic factors for the occurrence of complications, using the Fracture Risk Assessment Tool (FRAX) | Initial hospitalization
  Fracture risk prior to injury will be calculated with the Fracture Risk Assessment Tool [FRAX] (http://www.shef.ac.uk/FRAX/index.htm).
  Additionally, the fracture risk will be considered as a prognostic factor (in the absence of regular BMD measurements) for the analysis of complications.
Quality of reduction | one year
  The results of fracture reduction are assessed with the following clinical and radiological evaluations : Varus/valgus deformity, Endo-/exorotation deformity, Limb length.

CONTACTS AND LOCATIONS:
Overall Officials: Beate P. Hanson, MD, Study Director — AO Clinical Investigation and Documentation, Davos, Switzerland
Locations (3):
- Princess Alexandra Hospital, Woolloongabba, Queensland, Australia
- Switzerland (2):
  - Cantonal Hospital Chur, Chur
  - Cantonal Hospital Lucerne, Lucerne